CLINICAL TRIAL: NCT04776889
Title: The Prognosis of Lipid Reprogramming With the HMG-CoA Reductase Inhibitor, Rosuvastatin, in Castrated Egyptian Prostate Cancer Patients
Brief Title: The Prognosis of Lipid Reprogramming With Rosuvastatin, in Castrated Egyptian Prostate Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Riham Karkeet, Assistant lecturer, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB1901-30303
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer Metastatic
Keywords: Prostate cancer; Rosuvastatin; Castration/Androgen deprivation; HMG-CoA Reductase; Lipid metabolism/; Survival; Aldoketoreductase 1C4; Prostate specific antigen; Alkaline phosphatase; Caveolin-1; ABCA-1; SLDL-RP1; Lipid profile; epidermal growth factor receptor
MeSH Terms: conditions — Prostatic Neoplasms; Hypoalphalipoproteinemias | interventions — Rosuvastatin Calcium; Castration

STUDY DESIGN:
Intervention Model Description: A cohort of 70 newly diagnosed metastatic prostate cancer patients were recruited. Blood samples were withdrawn from all patients at baseline to monitor parameters under investigation. Then, all patients were subjected to surgical castration and divided in to two groups. Group I included 30 patients and served as control (statin non-users). Group II included 40 patients treated with Rosuvastatin (20 mg/day) for 6 months and served as statin users.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control/statin non-users (Active Comparator): newly diagnosed metastatic prostate cancer patients who underwent surgical castration in the form of bilateral subcapsular orchiectomy.
  Interventions: Procedure: surgical castration
- Interventional/statin users (Experimental): newly diagnosed metastatic prostate cancer patients who underwent surgical castration in the form of bilateral subcapsular orchiectomy and administered rosuvastatin 20 mg/day for 6 months
  Interventions: Drug: Rosuvastatin 20mg

INTERVENTIONS:
Drug: Rosuvastatin 20mg — Rosuvastatin 20mg/day for 6 months added to bilateral subcapsular orchiectomy
  Arms: Interventional/statin users
Procedure: surgical castration — bilateral subcapsular orchiectomy
  Arms: Control/statin non-users

SUMMARY:
Aim: The role of surgical castration and rosuvastatin treatment on lipid profile and lipid metabolism related markers was evaluated for their prognostic significance in metastatic prostate cancer (mPC) patients.

Methods: A total of 70 newly diagnosed castrated mPC patients treated with castration were recruited and divided into two groups: Group I included 30 patients and served as control (statin non-users) while group II included 40 patients treated with Rosuvastatin (20 mg/day) for 6 months and served as statin users. Prostate specific antigen (PSA), epidermal growth factor receptor (EGFR), Caveolin-1, lipid profile (LDL, HDL, triglycerides and cholesterol) and lipid metabolism related markers (aldoketoreductase (AKR1C4), HMGCoA reductase, ABCA1, and SLDL RP1) were measured at baseline, after 3 and 6 months. Overall survival (OS) were analyzed by Kaplan-Meier and COX regression for prognostic significance.

DETAILED DESCRIPTION:
This prospective randomized controlled study was conducted at the National Cancer Institute (NCI), Cairo University. The study ID BB1901-30303 was approved by the Institutional Human Research Ethics Committee of NCI, Egypt, Number 00004025, with IRB review Number 201819019.3 and conducted in accordance with the Declaration of Helsinki with informed consent was taken from all participants. The study included 70 Egyptian metastatic prostate cancer (m PC) patients who were treated and followed up in the NCI hospital in the period from January 2019 till December 2020. Patients were recruited from January to June 2019, then followed-up to December 2020.

Blood samples were withdrawn from all patients at baseline to monitor parameters under investigation. Then, all patients were subjected to surgical castration and divided in to two groups. Group I included 30 patients and served as control (statin non-users). Group II included 40 patients treated with Rosuvastatin (20 mg/day) for 6 months and served as statin users. Then, blood samples were withdrawn from the two groups after 3 and 6 months. Full demographic information and clinicopatholologic characteristics were obtained for each patient including; age, comorbid diseases, initial complain symptoms, family history of malignancy, smoking status and performance status. Also, serum level of prostate specific antigen (PSA) and alkaline phosphatase (ALP), Gleason score and metastasis sites were recorded. The treatment modality and decision making were according to NCI guidelines.

Collected whole blood samples into k.EDTA tubes were incubated at room temperature for 15 minutes and then centrifuged for 20 minutes at 1500 rpm. The plasma supernatant was carefully collected and freezed until analysis. Plasma protein concentrations of some lipid reprogramming and prostate cancer aggressiveness markers were measured. Kits were probed against human soluble low density lipoprotein receptor related protein -1 (SLDLRP-1; catalogue number: SL2705Hu), human ATP binding cassette transporter A-1 (ABCA-1; catalogue number: SL0314Hu), Human Aldoketo-reductase family 1 member C4 (AKR-1C4; catalogue number: SL3032Hu), human 3-hydroxy-3-methylglutaryl Co-enzyme A reductase (HMGCR; catalogue number: SL3030Hu), human epidermal growth factor receptor (EGFR; catalogue number: SL0665Hu) and human Caveolin-1 (Cav-1; catalogue number: SL0427Hu). Procedures were carried out in accordance with the manufacturer's instructions. The concentration of the markers in plasma samples was calculated by comparing the OD of the samples to the corresponding plotted standard curves.

Data management and statistical analysis were performed using The Statistical Package for Social Sciences (SPSS) version 24. Normal distribution and variance homogeneity of data were assessed using the Kolmogorov-Smirnov and Levene's tests, respectively. Numerical data were summarized using median and interquartile range (IQR). Categorical data were summarized as count and percentage. Patients were stratified according to their clinicopathological factors and for more than two subgroups of patients, the change in measured parameters were tested for significance using Kruskal-Wallis test and the pairwise comparison were done using Mann-Whitney. The change in proteins concentration over time was tested using Friedman test of significance. Spearman correlation analysis was used to test all possible correlations. Kaplan- Meier survival analysis was used to calculate the cumulative survival rate as well as median levels of OS after two years of follow up. OS was calculated from date of diagnosis to date of death by any cause. Living patients or patients lost to follow-up were censored on the last known alive date. The hazardous effect of death or progression Cox proportion hazard Model was used to evaluate the hazardous effect of different clinicopathological and proteins levels on death and progression. All P-values are two-sided. P-values < 0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Naïve newly diagnosed with metastatic prostate cancer
* Age ≥ 50 years.
* No psychological or geographical barriers for regular follow up of the patients.

Exclusion Criteria:

* Age < 50 years.
* psychological or geographical barriers for regular follow up of the patients.

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Lipid profile | 6 months
  effect of adding rosuvastatin to surgical castration on the lipid profile (LDL, triglycerides, cholesterol, HDL) in mg/dl
Aggressiveness parameters | 6 months
  effect of adding rosuvastatin to surgical castration on the PSA in ng/ml
Aggressiveness parameters | 6 months
  effect of adding rosuvastatin to surgical castration on the ALP in IU/L
Aggressiveness parameters | 6 months
  effect of adding rosuvastatin to surgical castration on the EGFR in ng/ml
Aggressiveness parameters | 6 months
  effect of adding rosuvastatin to surgical castration on the Caveolin-1 in pg/ml
Lipid metabolism parameters | 6 months
  effect of adding rosuvastatin to surgical castration on HMG-CoA reductase in ng/ml
Lipid metabolism parameters | 6 months
  effect of adding rosuvastatin to surgical castration on SLDLRP1 in pg/ml
Lipid metabolism parameters | 6 months
  effect of adding rosuvastatin to surgical castration on AKR1C4 ng/L
Lipid metabolism parameters | 6 months
  effect of adding rosuvastatin to surgical castration on ABCA-1 in pg/ml

SECONDARY OUTCOMES:
short-term clinical outcome | 18 months
  disease progression/regression
short-term clinical outcome | 18 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
requests for individual participant data should be directed to riham.karkeet@nci.cu.edu.eg, and shall not be limited to specific institutes/researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: for 2 years after publication
Access Criteria: requests for participant data should be directed to riham.karkeet@nci.cu.edu.eg, and shall not be limited to specific institutes/researchers

REFERENCES:
- [Derived] Karkeet RM, Zekri AN, Sayed-Ahmed MM, Sherif GM, Salem SE, Abdelbary A, Fouad MA, Saad SY. The prognosis of lipid reprogramming with the HMG-CoA reductase inhibitor, rosuvastatin, in castrated Egyptian prostate cancer patients: Randomized trial. PLoS One. 2022 Dec 8;17(12):e0278282. doi: 10.1371/journal.pone.0278282. eCollection 2022. PMID 36480560